CLINICAL TRIAL: NCT05020392
Title: Efficacy and Safety of Autologous Cells Derived Anti-CD19 CAR-Engineered T Cells With Concurrent BTK Inhibitor for B Cell Lymphoma：a Single-center, Open-label, Pragmatic Clinical Trial
Brief Title: Autologous Cells Derived Anti-CD19 CAR-Engineered T Cells With Concurrent BTK Inhibitor for B Cell Lymphoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Wuhan Si'an Medical Technology Co., Ltd (Unknown)
Responsible Party: Principal Investigator, MEI HENG, Proferssor, Cheif Doctor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: auto-CART-CD19 cells and BTKi
Record Dates: First submitted 2021-08-19; First posted 2021-08-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Diffuse Large B Cell Lymphoma; Burkitt Lymphoma; Follicular Lymphoma; Chronic Lymphocytic Leukemia; Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Burkitt Lymphoma; Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell

STUDY DESIGN:
Intervention Model Description: This study was a pragmatic clinical trial in which patients were divided into two groups, one receiving anti-CD19 CAR-T cells infusion, the other group receiving anti-CD19 CAR-T cells infusion and concurrent oral BTK inhibitor.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Effective of CAR-T-CD19 cells with concurrent BTK inhibitor (Experimental): After enrollment, all subjects will receive oral BTK inhibitor immediately and BTK inhibitor treatment will continue for up to 90 days (or longer for who are benefiting from BTK inhibitor) after CAR-T-CD19 infusion. Eligible patients will undergo leukapheresis to obtain peripheral blood mononuclear cells (PBMCs) for CAR T-cell production. Upon successful generation CAR-T-CD19 product, participants will receive fludarabine-based lymphodepletion chemotherapy, followed by infusion of CAR-T-CD19 cells (2*10^6 cells/kg) on day 0 and day 1 respectively.
  Interventions: Drug: BTK inhibitor+ Fludarabine-based chemotherapy + CAR-T-CD19 Cells
- Effective of CAR-T-CD19 cells monotherapy (Active Comparator): Eligible patients will undergo leukapheresis to obtain peripheral blood mononuclear cells (PBMCs) for CAR T-cell production. Upon successful generation CAR-T-CD19 product, participants will receive fludarabine-based lymphodepletion chemotherapy, followed by infusion of CAR-T-CD19 cells (2*10^6 cells/kg) on day 0 and day 1 respectively.
  Interventions: Drug: Fludarabine-based chemotherapy + CAR-T-CD19 Cells

INTERVENTIONS:
Drug: BTK inhibitor+ Fludarabine-based chemotherapy + CAR-T-CD19 Cells — BTK inhibitor from enrollment to more than 90 days after CAR-T-CD19 infusion. Fludarabine-based lymphodepletion chemotherapy was followed by CART19 infusion at a dose of 1x10^6/kg on day 0 and day 1 respectively.
  Arms: Effective of CAR-T-CD19 cells with concurrent BTK inhibitor
Drug: Fludarabine-based chemotherapy + CAR-T-CD19 Cells — Fludarabine-based lymphodepletion chemotherapy was followed by CART19 infusion at a dose of 1x10^6/kg on day 0 and day 1 respectively.
  Arms: Effective of CAR-T-CD19 cells monotherapy

SUMMARY:
This is a single-center, open-label and pragmatic clinical trial to evaluate the primary efficacy and safety of anti-CD19 chimeric antigen receptor (CAR)-modified T cells (CART-CD19) with concurrent BTK inhibitor in patients with relapsed or refractory B cell lymphoma

DETAILED DESCRIPTION:
Anti-CD19 chimeric antigen receptor (CAR) T-cell has shown dramatical efficacy in B cell malignancies. And Bruton tyrosine kinase (BTK) inhibitor agents have been validated as an effective drug to treat B cell malignancies. Combined therapies comprising ibrutinib (a BTK inhibitor) and anti-CD19 CAR-T cells in patients with CLL after ibrutinib failure are considered feasible and safe.

Ibrutinib is the first-generation BTK inhibitror and Zanubrutinib is the second-generation BTK inhibitor. Orelabrutinib is a newly developed BTK inhibitor with high selectivity and have received its approval in China. Autologous cells derived T cells are purified and transduced with a lentiviral vector encoding the humanized CD19 scFv.

To evaluate whether the addition of BTK inhibitor (Ibrutinib, Zanubrutinib and Orelabrutinib) in anti-CD19 CAR-T cells therapy would further improve efficacy and safety, we intend to conduct this pragmatic clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years and ≤70 years.
2. Expected survival over 6 months.
3. Eastern Cooperative Oncology Group score≤ 2.
4. Diagnosed pathologically and histologically CD19+B cell lymphoma, including mantle cell lymphoma, chronic lymphocytic leukemia, follicular cell lymphoma, Burkitt lymphoma and diffuse large B cell lymphoma.
5. Patients have failed at least 1 line of prior therapy
6. Negativity of blood pregnancy test for woman, and participants use effective methods of contraception until last follow-up.
7. Patient or his or her legal guardian voluntarily participates in and signs an informed consent form.

   -

Exclusion Criteria:

1. Investigators judge the patients with gastrointestinal lymph node and/or central nervous system involvement who may be at high-risk of receiving CAR-T-CD19 cell treatment.
2. Existing or preexisting CNS conditions, such as epileptic seizures, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any CNS related autoimmune diseases.
3. Patients with graft-versus-host reaction and need immunosuppressive agents, or patients with autoimmune diseases.
4. Participants with other active malignancies (except non-melanoma skin cancer and cervical cancer) within five years.
5. History of Richter's syndrome.
6. History of any one of the following cardiovascular conditions within the past 6 months: Class III or IV heart failure as defined by the New York Heart Association (NYHA), cardiac angioplasty or stenting, myocardial infarction, unstable angina, or other clinically significant cardiac disease.
7. Patients who are pregnant or breast-feeding.
8. Patients with any one of the following terms:

   A. Creatine >2.5mg/dl (221.0umol/L). B. Alanine aminotransferase/aspartate aminotransferase >3 times the upper limit of normal (ULN).

   C. Total bilirubin>2.0 mg/dl (34.2umol/L).
9. Major surgery within 4 weeks of randomization.
10. Systemic steroids are used within 2 weeks before apheresis (Except for those who are using inhaled steroids recently or currently).
11. Patients receive cytotoxic chemotherapy or radiotherapy within 21 days before enrollment (Tyrosine kinase inhibitors or other targeted therapies can be used two weeks before lymphodepleting chemotherapy).
12. Prior treatment with any gene therapy product.
13. Active hepatitis B, active hepatitis C, or active human immunodeficiency virus (HIV) infection.
14. Systemic fungal, bacterial, viral, or other infection that is not controlled.
15. The absolute value of lymphocytes was too low to manufacture CAR-T cells.
16. Other conditions considered inappropriate by the researcher.

    -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-09-14 (Actual); Primary Completion 2023-10-13 (Estimated); Study Completion 2024-10-13 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-related Adverse Events | within 2 years after infusion
  Therapy-related adverse events (AE), including severe adverse events (SAE) and laboratory outliers with clinical significance, will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0).

SECONDARY OUTCOMES:
Overall response rate (ORR) of administering CAR-T-CD19 cells or CAR-T-CD19 cells with oral BTK inhibitor in Relapsed/Refractory B cell lymphoma. | within 2 years after infusion
  ORR will be assessed from CAR-T cell infusion to death or last follow-up (censored).
Duration of Response (DOR) of administering CAR- T-CD19 cells or CAR-T-CD19 cells with oral BTK inhibitor in Relapsed/Refractory CD19+ B-cell lymphoma. | within 2 years after infusion
  DOR will be assessed from CAR-T cell infusion to death or last follow-up (censored).
Overall survival (OS) of administering CAR- T-CD19 cells or CAR-T-CD19 cells with oral BTK inhibitor in Relapsed/Refractory CD19+ B-cell lymphoma. | within 2 years after infusion
  OS will be assessed from CAR-T cell infusion to death or last follow-up (censored).
PFS will be assessed from CAR-T cell infusion to death or last follow-up | within 2 years after infusion
  Progress-free survival (PFS) of administering CAR- T-CD19 cells or CAR-T-CD19 cells with oral BTK inhibitor in Relapsed/Refractory CD19+ B-cell lymphoma.
Complete response rate (CR) of administering CAR-T-CD19 cells or CAR-T-CD19 cells with oral BTK inhibitor in Relapsed/Refractory B cell lymphoma. | within 2 years after infusion
  CR will be assessed from CAR-T cell infusion to death or last follow-up (censored).
Partial response rate (PR) of administering CAR-T-CD19 cells or CAR-T-CD19 cells with oral BTK inhibitor in Relapsed/Refractory B cell lymphoma. | within 2 years after infusion
  PR will be assessed from CAR-T cell infusion to death or last follow-up.

OTHER OUTCOMES:
In vivo expansion and survival of CAR-T-CD19 cells | within 2 years after infusion
  Quantity of CAR-T-CD19 CAR copies in bone marrow, peripheral blood and cerebrospinal fluid will be determined by using quantitative polymerase chain reaction.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Hu, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gauthier J, Hirayama AV, Purushe J, Hay KA, Lymp J, Li DH, Yeung CCS, Sheih A, Pender BS, Hawkins RM, Vakil A, Phi TD, Steinmetz RN, Shadman M, Riddell SR, Maloney DG, Turtle CJ. Feasibility and efficacy of CD19-targeted CAR T cells with concurrent ibrutinib for CLL after ibrutinib failure. Blood. 2020 May 7;135(19):1650-1660. doi: 10.1182/blood.2019002936. PMID 32076701
- [Background] Fraietta JA, Beckwith KA, Patel PR, Ruella M, Zheng Z, Barrett DM, Lacey SF, Melenhorst JJ, McGettigan SE, Cook DR, Zhang C, Xu J, Do P, Hulitt J, Kudchodkar SB, Cogdill AP, Gill S, Porter DL, Woyach JA, Long M, Johnson AJ, Maddocks K, Muthusamy N, Levine BL, June CH, Byrd JC, Maus MV. Ibrutinib enhances chimeric antigen receptor T-cell engraftment and efficacy in leukemia. Blood. 2016 Mar 3;127(9):1117-27. doi: 10.1182/blood-2015-11-679134. Epub 2016 Jan 26. PMID 26813675
- [Background] Cameron F, Sanford M. Ibrutinib: first global approval. Drugs. 2014 Feb;74(2):263-71. doi: 10.1007/s40265-014-0178-8. PMID 24464309
- [Derived] Luo W, Zhang Y, Li C, Xu J, Wu Z, Wang X, Kang Y, Liao D, Kou H, Xie W, Xiong W, Deng J, Mei H, Hu Y. BTK Inhibitor Synergizes With CD19-Targeted Chimeric Antigen Receptor-T Cells in Patients With Relapsed or Refractory B-Cell Lymphoma: An Open-Label Pragmatic Clinical Trial. Cancer Med. 2025 Oct;14(20):e71321. doi: 10.1002/cam4.71321. PMID 41123227